CLINICAL TRIAL: NCT03014596
Title: What Matters to You? How to Strengthen Adolescent User Involvement in Primary Mental Health Services With Systematic Idiographic Assessment
Brief Title: What Matters to You?
Acronym: Assert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionsenter for barn og unges psykiske helse (Other)
Collaborators: Norwegian Extra Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Simon-Peter Neumer, PhD, Regionsenter for barn og unges psykiske helse
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016/FO77493
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Behavioural, Emotional, and Psychosocial Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Assert-method will be used in the counselling of adolescents with mental health problems
  Interventions: Other: Assert
- Control (No Intervention): Treatment as usual, i.e. tha Assert-method will not be used in the counselling

INTERVENTIONS:
Other: Assert — The Assert-method is a counselling method used to assess and systematically follow up the individual adolescents' perceived needs.
  Arms: Intervention

SUMMARY:
Procedures for systematic user involvement in primary mental health services are lacking, and several adolescents are dissatisfied with their opportunities to influence the service provided. The research on the effects of user involvement is scarce, especially regarding user involvement for children and adolescents. Hence, we suggest introducing an idiographic assessment tool in a selection of Norwegian primary mental health services. Idiographic assessment is a way of measuring psychological constructs, by using tools specifically adapted for each individual respondent.

This protocol describes the implementation and evaluation of a user involvement tool called 'Assert', in Norwegian primary mental health services. Assert is a simple tool where the adolescents themselves decide the goals or themes that they would like to address in collaboration with their service provider. Assert is scored each time the adolescent and the service provider meet, to monitor progress toward the goal. A randomised controlled trial design is proposed for this study. Assert will be implemented in 5-10 Norwegian municipalities, and will include 250 participants between 12 and 23 years. The objective of the study is to examine the relationship between Assert and perceived user involvement. Are idiographic measures an adequate way to operationalise user involvement on an individual level? And if so, can user involvement (i.e. Assert) have an effect on quality of life and mental health in adolescents? And lastly qualitative analyses of the adolescents' themes and goals will be conducted to explore what matters to the adolescents that visit primary mental health services in Norwegian municipalities.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 12 and 23 years, with behavioural, emotional, and psychosocial problems

Exclusion Criteria:

* severe psychopathological disorders
* severe drug addiction
* intellectual disabilities

Ages: 12 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Strengths and difficulties questionnaire (SDQ) | One year
Inventory of Life Quality in Children and Adolescents (ILC) | One year
Multidimensional Health Locus of Control (MHLC) | One year

SECONDARY OUTCOMES:
The Assert measurement tool | One year
  An ideographic assessment and monitoring tool, used as a part of the Assert method
User involvement questionnaire | One year
  Perceived degree of user involvement

CONTACTS AND LOCATIONS:
Overall Officials: Turid Suzanne Berg-Nielsen, PhD, Principal Investigator — Regional Centre for Child and Adolescent Mental Health, Eastern and Southern Norway (RBUP)
Locations (11):
- Norway (11):
  - Ål kommune, Ål
  - Ringerike kommune, Hønefoss
  - Kongsberg kommune, Kongsberg
  - Skedsmo kommune, Lillestrøm
  - Lørenskog kommune, Lørenskog
  - Eidsberg Kommune, Mysen
  - Bydel Søndre Nordstrand, Oslo
  - UngArena, Oslo
  - Familiehuset Adler, Tønsberg
  - Nome kommune, Ulefoss
  - Våler kommune, Våler

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tollefsen TK, Neumer SP, Berg-Nielsen TS. "What matters to you?": A randomized controlled effectiveness trial, Using Systematic Idiographic Assessment as an intervention to Increase Adolescents' perceived control of their mental health. J Adolesc. 2020 Jan;78:53-61. doi: 10.1016/j.adolescence.2019.11.006. Epub 2019 Dec 10. PMID 31835096